CLINICAL TRIAL: NCT04429932
Title: An Open-Label, Randomized, Crossover Study to Assess Nicotine Uptake, Tobacco-Related Biomarkers of Exposure, Biomarkers of Potential Harm, and Puff Topography With Use of mybluTM Electronic Cigarettes in Adult Smokers
Brief Title: A Study to Evaluate Nicotine Uptake and Biomarkers in Adult Smokers Using mybluTM Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fontem US LLC (Industry)
Collaborators: Fontem Ventures BV (Industry)
Responsible Party: Sponsor
Organization: Fontem Ventures BV (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CA22736
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Product use sequence ABDC (Experimental): Subjects use MybluTM e-cigarette product variant A (2.4% nicotine) ad libitum for 2 days, then switch to use variant B (2.4% nicotine) for 2 days, then D (2.4% nicotine) for 2 days and then C (2.4% nicotine) for 2 days. A washout period of 12 hours product abstinence is observed between product variants. For each product variant, in the morning of the second product use day, a controlled product use session is performed (10 puffs taken at 30-second intervals, with puffs 3 seconds in duration).
  Interventions: Other: Myblu flavor A_2.4; Other: Myblu flavor B_2.4; Other: Myblu flavor C_2.4; Other: Myblu flavor D_2.4
- Product use sequence BCAD (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu flavor A_2.4; Other: Myblu flavor B_2.4; Other: Myblu flavor C_2.4; Other: Myblu flavor D_2.4
- Product use sequence CDBA (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu flavor A_2.4; Other: Myblu flavor C_2.4; Other: Myblu flavor D_2.4
- Product use sequence DACB (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu flavor A_2.4; Other: Myblu flavor B_2.4; Other: Myblu flavor C_2.4; Other: Myblu flavor D_2.4
- Product use sequence EFHG (Experimental): Subjects use MybluTM e-cigarette product variant E (1.2% nicotine) ad libitum for 2 days, then switch to use variant F (1.2% nicotine) for 2 days, then H (2.4% nicotine) for 2 days and then G (2.4% nicotine) for 2 days. A washout period of 12 hours product abstinence is observed between product variants. For each product variant, in the morning of the second product use day, a controlled product use session is performed (10 puffs taken at 30-second intervals, with puffs 3 seconds in duration).
  Interventions: Other: Myblu flavor E_1.2; Other: Myblu flavor F_1.2; Other: Myblu flavor G_2.4; Other: Myblu flavor H_2.4
- Product use sequence FGEH (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu flavor E_1.2; Other: Myblu flavor F_1.2; Other: Myblu flavor G_2.4; Other: Myblu flavor H_2.4
- Product use sequence GHFE (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu flavor E_1.2; Other: Myblu flavor F_1.2; Other: Myblu flavor G_2.4; Other: Myblu flavor H_2.4
- Product use sequence HEGF (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu flavor E_1.2; Other: Myblu flavor F_1.2; Other: Myblu flavor G_2.4; Other: Myblu flavor H_2.4

INTERVENTIONS:
Other: Myblu flavor A_2.4 — Use of Myblu e-cigarette with flavor 1 at 2.4% nicotine
  Arms: Product use sequence ABDC; Product use sequence BCAD; Product use sequence CDBA; Product use sequence DACB
Other: Myblu flavor B_2.4 — Use of Myblu e-cigarette with flavor 2 at 2.4% nicotine
  Arms: Product use sequence ABDC; Product use sequence BCAD; Product use sequence DACB
Other: Myblu flavor C_2.4 — Use of Myblu e-cigarette with flavor C at 2.4% nicotine
  Arms: Product use sequence ABDC; Product use sequence BCAD; Product use sequence CDBA; Product use sequence DACB
Other: Myblu flavor D_2.4 — Use of Myblu e-cigarette with flavor D at 2.4% nicotine
  Arms: Product use sequence ABDC; Product use sequence BCAD; Product use sequence CDBA; Product use sequence DACB
Other: Myblu flavor E_1.2 — Use of Myblu e-cigarette with flavor 1 at 1.2% nicotine
  Arms: Product use sequence EFHG; Product use sequence FGEH; Product use sequence GHFE; Product use sequence HEGF
Other: Myblu flavor F_1.2 — Fse of Myblu e-cigarette with flavor F at 1.2% nicotine
  Arms: Product use sequence EFHG; Product use sequence FGEH; Product use sequence GHFE; Product use sequence HEGF
Other: Myblu flavor G_2.4 — Use of Myblu e-cigarette with flavor G at 2.4% nicotine
  Arms: Product use sequence EFHG; Product use sequence FGEH; Product use sequence GHFE; Product use sequence HEGF
Other: Myblu flavor H_2.4 — Use of Myblu e-cigarette with flavor H at 2.4% nicotine
  Arms: Product use sequence EFHG; Product use sequence FGEH; Product use sequence GHFE; Product use sequence HEGF

SUMMARY:
This study evaluates the overall performance of the currently-marketed MybluTM e-cigarette device and pods, as assessed by nicotine uptake, exposure to smoke constituents, safety and consumer satisfaction, over 8 days. The study is designed as an open-label, randomized study in adult smokers.

Subjects are invited to participate to a second part of the study, for 5 additional days, to compare the use of MybluTM to the use of subject's usual brand combustible cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* smoking an average of at least 10 manufactured combustible cigarettes per day for at least 12 months prior to Screening
* tested positive for urine cotinine (≥ 200 ng/mL) at Screening
* exhaled carbon monoxide > 10 ppm (parts per million) at Screening

Exclusion Criteria:

* relevant illness history
* relevant medication use
* body mass index (BMI) > 40 kg/m2 or < 18 kg/m2 at Screening
* allergy to propylene glycol or glycerin
* use of nicotine-containing products other than manufactured combustible cigarettes within 14 days prior to Check-in
* use of any prescription smoking cessation treatments within 3 months prior to Check-in
* smokers who draw smoke from the cigarette into the mouth and throat but do not inhale
* planning to quit smoking during the study
* female subjects who are pregnant, lactating, or intend to become pregnant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Morris P, McDermott S, Chapman F, Verron T, Cahours X, Stevenson M, Thompson J, Chaudhary N, O'Connell G. Reductions in biomarkers of exposure to selected harmful and potentially harmful constituents following exclusive and partial switching from combustible cigarettes to myblu electronic nicotine delivery systems (ENDS). Intern Emerg Med. 2022 Mar;17(2):397-410. doi: 10.1007/s11739-021-02813-w. Epub 2021 Aug 26. PMID 34435305

RESULTS

PARTICIPANT FLOW:
Groups:
- Product Use Sequence ABDC: Subjects use MybluTM e-cigarette product variant A (2.4% nicotine) ad libitum for 2 days, then switch to use variant B (2.4% nicotine) for 2 days, then D (2.4% nicotine) for 2 days and then C (2.4% nicotine) for 2 days. A 12-hour washout period is observed between product variants. For each product variant, in the morning of the second product use day, a controlled product use session is performed (10 puffs taken at 30-second intervals, with puffs 3 seconds in duration).
  Myblu flavor A_2.4: Use of Myblu e-cigarette with flavor 1 at 2.4% nicotine
  Myblu flavor B_2.4: Use of Myblu e-cigarette with flavor 2 at 2.4% nicotine
  Myblu flavor C_2.4: Use of Myblu e-cigarette with flavor C at 2.4% nicotine
  Myblu flavor D_2.4: Use of Myblu e-cigarette with flavor D at 2.4% nicotine
- Product Use Sequence EFHG: Subjects use MybluTM e-cigarette product variant E (1.2% nicotine) ad libitum for 2 days, then switch to use variant F (1.2% nicotine) for 2 days, then H (2.4% nicotine) for 2 days and then G (2.4% nicotine) for 2 days. A 12-hour washout period is observed between product variants. For each product variant, in the morning of the second product use day, a controlled product use session is performed (10 puffs taken at 30-second intervals, with puffs 3 seconds in duration).
  Myblu flavor E_1.2: Use of Myblu e-cigarette with flavor 1 at 1.2% nicotine
  Myblu flavor F_1.2: Fse of Myblu e-cigarette with flavor F at 1.2% nicotine
  Myblu flavor G_2.4: Use of Myblu e-cigarette with flavor G at 2.4% nicotine
  Myblu flavor H_2.4: Use of Myblu e-cigarette with flavor H at 2.4% nicotine
Period: Overall Study
Arm/Group | Product Use Sequence ABDC | Product Use Sequence BCAD | Product Use Sequence CDBA | Product Use Sequence DACB | Product Use Sequence EFHG | Product Use Sequence FGEH | Product Use Sequence GHFE | Product Use Sequence HEGF
Started | 4 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Completed | 3 | 5 | 5 | 2 | 5 | 5 | 5 | 5
Not Completed | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Product Use Sequence ABDC | Product Use Sequence BCAD | Product Use Sequence CDBA | Product Use Sequence DACB | Product Use Sequence EFHG | Product Use Sequence FGEH | Product Use Sequence GHFE | Product Use Sequence HEGF | Total
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (15.8) | 49.0 (4.9) | 38.0 (9.2) | 32.6 (7.2) | 36.4 (7.0) | 40.8 (8.7) | 46.4 (10.0) | 50.0 (6.4) | 41.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 2 | 2 | 3 | 3 | 14
  Male | 3 | 4 | 4 | 4 | 3 | 3 | 2 | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 3 | 1 | 0 | 1 | 0 | 9
  Not Hispanic or Latino | 3 | 4 | 3 | 2 | 4 | 5 | 4 | 5 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.8 (4.2) | 30.5 (5.5) | 28.2 (5.0) | 26.1 (4.1) | 29.4 (4.4) | 29.7 (7.7) | 28.5 (4.2) | 28.7 (6.3) | 28.4 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Nicotine Concentration in Blood
Description: Maximum nicotine concentration in blood (Cmax)
Time Frame: 180 minutes following the start of the controlled product use session on Day 2 (12 measurements over the period)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Product Variant A: MyBlu e-cigarette variant A (2.4% nicotine)
- Product Variant B: MyBlu e- igarette variant B (2.4% nicotine)
- Product Variant C: MyBlu e-cigarette variant C (2.4% nicotine)
- Product Variant D: MyBlu e-cigarette variant D (2.4% nicotine)
- Product Variant E: MyBlu e- cigarette variant E (1.2% nicotine)
- Product Variant F: MyBlu e-cigarette variant F (1.2% nicotine)
- Product Variant G: MyBlu e-cigarette variant G (2.4% nicotine)
- Product Variant H: MyBlu e-cigarette variant H (2.4% nicotine)
Arm/Group | Product Variant A | Product Variant B | Product Variant C | Product Variant D | Product Variant E | Product Variant F | Product Variant G | Product Variant H
Number analyzed (Participants) | 14 | 14 | 15 | 17 | 20 | 20 | 20 | 20
ng/mL | 6.6 (137.5) | 7.9 (91.8) | 5.6 (107.2) | 6.0 (184.5) | 2.6 (88.7) | 2.7 (91.4) | 4.4 (94.4) | 3.5 (295.6)

2. Primary Outcome: Concentration of Carboxyhemoglobin in Blood
Description: Change from baseline in the concentration of carboxyhemoglobin (COHb) in whole blood.
Time Frame: Baseline and 8 days
Population: Data is missing for 3 participants at the 8 days timepoint
Measure: Mean (Standard Deviation); unit: % saturation
Groups:
- Exclusive MyBlu E-cigarette Use: Subjects who used any MyBlu e-cigarette variant for 8 days (all subjects who completed Part 1 of the study)
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 38
% saturation
  Baseline value | 5.4 (1.8)
  Change from baseline: number analyzed (Participants) | 35
  Change from baseline | -4.0 (1.8)

3. Primary Outcome: Amount of 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol in Urine in 24 Hours
Description: Change from baseline in the amount of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL), a biomarker of exposure to 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK), excreted in urine during 24 hours (creatinine adjusted).
Time Frame: Baseline and 8 days
Population: Data is missing for 3 participants at the 8 days timepoint
Measure: Mean (Standard Deviation); unit: ng/g creatinine
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 38
ng/g creatinine
  Baseline value | 176.2 (87.4)
  Change from baseline | -134.8 (66.5)

4. Primary Outcome: Amount of 3-hydroxypropylmercapturic Acid in Urine in 24 Hours
Description: Change from baseline in the amount of 3-hydroxypropylmercapturic acid (3-HPMA), a biomarker of exposure to acrolein, excreted in urine during 24 hours (creatinine adjusted).
Time Frame: Baseline and 8 days
Population: Data is missing for 3 participants at the 8 days timepoint
Measure: Mean (Standard Deviation); unit: ug/g creatinine
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 38
ug/g creatinine
  Baseline value | 756.2 (279.3)
  Change from baseline: number analyzed (Participants) | 35
  Change from baseline | -599.3 (276.6)

5. Primary Outcome: Amount of S-phenyl Mercapturic Acid in Urine in 24 Hours
Description: Change from baseline in the amount of S-phenyl mercapturic acid (S-PMA), a biomarker of exposure to benzene, excreted in urine during 24 hours (creatinine adjusted).
Time Frame: Baseline and 8 days
Population: Data is missing for 3 participants at the 8 days timepoint
Measure: Mean (Standard Deviation); unit: ug/g creatinine
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 38
ug/g creatinine
  Baseline value | 2.6 (1.4)
  Change from baseline: number analyzed (Participants) | 35
  Change from baseline | -2.5 (1.4)

6. Secondary Outcome: Level of White Blood Cells
Description: The change from baseline in the level of white blood cells, a biomarker of potential harm.
Time Frame: Baseline and 8 days
Population: Data is missing for 3 participants at the 8 days timepoint
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 38
cells*10^9/L
  Baseline value | 6.9 (1.5)
  Change from baseline: number analyzed (Participants) | 35
  Change from baseline | -0.6 (1.0)

7. Secondary Outcome: Spirometry: Forced Expiratory Volume in 1 Second
Description: The percent-predicted forced expiratory volume in 1 second (FEV1) measurement conducted in accordance with the 2005 American Thoracic Society / European Respiratory Society Joint Task Force on the standardization of spirometry, with subject in a sitting position following at least 15 minutes of rest and at least 1 hour from the last product use.
Time Frame: Baseline and 8 days
Population: Data is missing for 3 participants at the 8 days timepoint
Measure: Mean (Standard Deviation); unit: Percent-predicted FEV1
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 38
Percent-predicted FEV1
  Baseline value | 98.0 (14.6)
  8 days timepoint | 98.6 (16.2)

8. Secondary Outcome: Spirometry: Forced Vital Capacity
Description: The percent-predicted forced vital capacity (FVC) measurement conducted in accordance with the 2005 American Thoracic Society / European Respiratory Society Joint Task Force on the standardization of spirometry, with subject in a sitting position following at least 15 minutes of rest and at least 1 hour from the last product use.
Time Frame: Baseline and 8 days
Population: Data is missing for 3 participants at the 8 days timepoint
Measure: Mean (Standard Deviation); unit: Percent-predicted FVC
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 38
Percent-predicted FVC
  Baseline value | 101.0 (14.6)
  8 days timepoint: number analyzed (Participants) | 35
  8 days timepoint | 100.3 (16.0)

9. Secondary Outcome: Subjective Measure: Urge to Smoke
Description: Urge to smoke score: Subjects answer the following question "How strong is your urge to smoke right now?" using a visual analogue scale. The scale ranges from "Not at all", given a score of 0, to "Extremely", given a score of 100, after ad libitum use of the product.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Product Variant A | Product Variant B | Product Variant C | Product Variant D | Product Variant E | Product Variant F | Product Variant G | Product Variant H
Number analyzed (Participants) | 16 | 15 | 14 | 17 | 20 | 20 | 20 | 20
score on a scale | 72.3 (21.9) | 76.4 (13.8) | 64.9 (23.4) | 67.6 (26.0) | 53.7 (32.6) | 54.4 (29.5) | 55.4 (29.9) | 59.0 (31.5)

ADVERSE EVENTS:
Time Frame: 9 days
Arm/Group | Product Variant A | Product Variant B | Product Variant C | Product Variant D | Product Variant E | Product Variant F | Product Variant G | Product Variant H
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/16 | 0/18 | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/16 | 0/18 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/18 | 1/16 | 1/16 | 1/18 | 2/20 | 1/20 | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Product Variant A (N=18) | Product Variant B (N=16) | Product Variant C (N=16) | Product Variant D (N=18) | Product Variant E (N=20) | Product Variant F (N=20) | Product Variant G (N=20) | Product Variant H (N=20)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contact dermitits (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT04429932/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT04429932/SAP_001.pdf